CLINICAL TRIAL: NCT01679990
Title: A Phase II, Randomized, Double-Blind, Multicenter, Multinational, Placebo-Controlled, Parallel- Groups Study to Evaluate the Safety and Efficacy of Intramuscular Injections of Allogeneic PLX-PAD Cells for the Treatment of Subjects With Intermittent Claudication (IC)
Brief Title: Safety and Efficacy of Allogeneic Cells for the Treatment of Intermittent Claudication(IC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pluristem Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PLX 1204-01
Record Dates: First submitted 2012-09-02; First posted 2012-09-06 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2017-01

CONDITIONS: Intermittent Claudication; Peripheral Artery Disease
MeSH Terms: conditions — Intermittent Claudication; Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (4):
- PLX-PAD Low dose (Experimental): PLX-PAD double low doses
  Interventions: Biological: PLX-PAD Low dose
- PLX-PAD high doses (Active Comparator): PLX-PAD double high dose
  Interventions: Biological: PLX-PAD high doses
- Placebo (Placebo Comparator): Double Placebo doses
  Interventions: Biological: Double Placebo
- PLX-PAD high dose +Placebo (Experimental): High dose+Placebo
  Interventions: Biological: high dose +Placebo

INTERVENTIONS:
Biological: PLX-PAD Low dose
  Arms: PLX-PAD Low dose
Biological: PLX-PAD high doses
  Arms: PLX-PAD high doses
Biological: Double Placebo
  Arms: Placebo
Biological: high dose +Placebo
  Arms: PLX-PAD high dose +Placebo

SUMMARY:
The objective of the study is to establish the safety profile of

Intramuscular PLX-PAD injections and to evaluate the clinical efficacy of it in IC subjects comprising of 4 treatment groups:

1. Double treatment of PLX-PAD low dose
2. Double treatment of PLX-PAD high dose
3. Double treatment of Placebo
4. Single treatment of PLX-PAD high dose and additional treatment of Placebo. Subjects will receive the assigned treatment twice to the affected leg, within 12-weeks interval between each treatment.

The study will be comprised of 5 stages:

Screening period of up to 4 weeks,first treatment of PLX-PAD or placebo followed by additional injection after 12 weeks and with follow-up of 12 months post second injection

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female subjects between 45 to 85 years of age (inclusive) at the time of screening visit.
* Subjects with a diagnosis of peripheral artery disease, secondary to atherosclerosis, confirmed by one of the following criteria assessed at the screening visit:

  * Resting ankle-brachial index (ABI) ≤ 0.80 or
  * Resting ABI ≤ 0.90 and >20% decrease in ABI from rest to exercise when measured within 1 minute after treadmill exercise or
  * Toe-brachial index (TBI) ≤ 0.60
* Lifestyle-limiting, moderate to severe claudication (symptoms present and stable for > 6 months and not significantly changed within the past 3 months prior to screening).
* Evidence of significant (>50%) stenosis infra-inguinal occlusive disease as confirmed by documented results from Duplex, MRA, CTA and/or contrast angiogram completed within 3 months prior to screening.
* The longest maximal walking distance (MWD) from the Screening Period exercise treadmill tests (ETT), utilizing a modified Gardner Protocol (Appendix I), must be between 1 and 10 minutes (inclusive).
* Subjects who have persistent claudication symptoms despite having been recommended an exercise program if feasible, and or despite having been on a stable dose of Cilostazol, if indicated. Subjects should be Cilostazol free for at least 2 weeks prior to the first ETT.
* Subjects should be receiving standard of care drugs for vascular disease including anti-platelet agent(s) and statin medication, as well as anti-hypertensive medication(s) and oral hypoglycemic agents/insulin, if indicated.
* Signed written informed consent.

Exclusion Criteria:

* Ischemic rest pain; ulceration or gangrene (Fontaine class III-IV; Rutherford category 4-6).
* Failed lower extremity arterial reconstruction (surgical or endovascular) or sympathectomy within the prior one month of screening.
* Planned revascularization (surgical or endovascular intervention) within 12 months after screening.
* Lower extremity arteries inflow obstruction (defined as a greater than 50% stenosis of aorta, iliac and/or common femoral arteries).
* History of Buerger's disease.
* Uncontrolled hypertension (defined as diastolic blood pressure > 100 mmHg or systolic blood pressure > 180 mmHg during screening).
* Uncontrolled diabetes defined as glucose control HbA1c > 9% at screening.
* Life-threatening ventricular arrhythmia - except in subjects with an implantable cardiac-defibrillator.
* Serum Creatinine level>2.5mg/dl.
* SGPT (ALT), SGOT (AST) >2.5 x upper limit of normal range.
* Hemoglobin < 10 g/dl.
* Unstable cardiovascular disease defined as myocardial infarction (STEMI or NSTEMI) within 3 months prior to screening, or unstable angina - characterized by increasingly frequent episodes with modest exertion or at rest, worsening severity, and prolonged episodes.
* Transient Ischemic Attack (TIA)/Stroke within 3 months prior to screening.
* Subjects with severe congestive heart failure symptoms (i.e. NYHA Stage III to IV).
* Subjects with Implant of mechanical prosthetic heart valve(s).
* Pulmonary disease requiring supplemental oxygen treatment on a daily basis.
* Severe, active infection of the involved extremity(ies), including osteomyelitis, fasciitis, or severe/purulent cellulitis.
* History of malignancy within 5 years prior screening requiring chemotherapy and/or radiotherapy and/or immunotherapy, excluding basal or squamous cell carcinoma of the skin.
* Exercise is limited by any condition other than IC, including but not limited to congestive heart failure, chronic pulmonary disease, angina pectoris, or degenerative joint disease.
* Uninterrupted use of warfarin or non-steroidal anti-inflammatory agents (with the exception of ibuprofen at doses up to 1,200 mg/day or Diclofenac at dose of 75mg/day).
* Subjects who are on oral anticoagulant therapy (warfarin, dabigatran, apixaban, endoxaban and rivaroxaban). Unless, upon primary care physician and/or Investigator's discretion the subjects who are on warfarin treatment can switch to Low Molecular Weight Heparin treatment (such as: Clexane) 5-7 days prior study treatment administration and return to warfarin treatment 24 hours post study treatment administration.
* Subjects who are taking immunosuppressive treatment (including high dose steroids).
* Known allergies to protein products (Bovine serum, or recombinant trypsin) used in the cell production process.
* Known sensitivity to Gentamycin.
* Known sensitivity to antihistamine drugs.
* History of hospitalization due to allergic/hypersensitivity reaction to any substance (e.g. Food or drug).
* Medical history of Human Immunodeficiency Virus (HIV) or syphilis positivity at time of screening.
* Known active Hepatitis B, or Hepatitis C infection at the time of screening.
* Pregnant or breast-feeding women or women of childbearing age not protected by an effective contraceptive method of birth control (such as double barrier, oral or parenteral hormonal, intrauterine device and spermicide).
* In the opinion of the Investigator, the subject is unsuitable for participating in the study.
* Subject is currently enrolled in, or has not yet completed a period of at least 30 days since ending other investigational device or drug trial(s).
* Subjects that have prior exposure to gene or cell based therapy.
* Subjects who are legally detained in an official institute.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2012-11-05; Primary Completion 2018-03-29 (Actual); Study Completion 2019-02-09 (Actual)

PRIMARY OUTCOMES:
Log ratio of week 52 maximal walking distance(MWD)to baseline MWD | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Denham, DO, Principal Investigator — Clinical Trials of Texas, Inc. 7940 Floyd Curl drive, Suite 700, San Antonio, Texas 78229; James Hampsey, MD, Principal Investigator — Tampa Bay Medical research, 3251 McMullen Booth Road, STE 303, Clearwater, FL 33761; Schulyer Jones, MD, Principal Investigator — Duke University,Durham, North Carolina, 27705, USA; Bret Weichmann, MD, Principal Investigator — Florida research Network, LLC 6800NW 9th Blvd Suite1, Gainesville, Florida 32605; Jeffrey W Olin, DO, Principal Investigator — Cardiovascular Institute, Mount Sinai School of Medicine , One Gustave L. Levy Place, New York, NY 10029; Alan T Hirsch, MD, Principal Investigator — Cardiovascular Division, MMC 508, University of Minnesota Medical school, Minneapolis, MN 55455; Sibu P. Saha, MD, Principal Investigator — University of Kentucky, Lexington, KY 40506-0057; David L Fried, MD, Principal Investigator — Omega Medical Research, Warwick, RI 02886; Berthold Amann, MD, Principal Investigator — Franziskus-Krankenhaus, Berlin Germany; Norbert Weiss, MD, Principal Investigator — Universitätsklinikum Carl Gustav Carus, Dresden, Germany; Sigrid Nikol, MD, Principal Investigator — ASKLEPIOS Klinik St. Georg, Hamburg Germany; Malcolm Foster, MD, Principal Investigator — Turkey Creek Medical Center, Knoxville TN 37934; Kathleen Cullen, MD, Principal Investigator — DMI Research, 6699 90th Ave. North, Pinellas Park FL; Mohler Emile, M.D, Principal Investigator — Hospital of the University of Pennsylvania, Philadelphia, PA 19104; Nadarajah Janaki, M.D, Principal Investigator — Aiyan Diabetes Center, Evans, GA 30809; Reuven Zimlichman, MD, Principal Investigator — Edith Wolfson Medical Center,62 HaLohamim Street, Holon, Israel; Changyoung Lim, MD, Principal Investigator — CHA Bundang Medical Center, CHA University, 59 Yatap-ro Bundang-Gu, Seongnam-Si, Gyeonggi-do 463-712, Korea; Weonyong Lee, MD, Principal Investigator — Hallym University Sacred Heart Hospital 22, Gwanpyeong-ro 170beon-gil, Dongan-gu, Anyang-si, Gyeonggi-do, 431-796, Korea; Sungwon Chung, MD, Principal Investigator — Pusan National University Hospital 179 Gudeok-Ro Seo-Gu, Busan, 602-739, Korea; Yousun Hong, MD, Principal Investigator — Ajou University School of Medicine; Jaeseung Shin, MD, Principal Investigator — Korea University; Kwangjo Cho, MD, Principal Investigator — Dong-A University Hospital; Dokyun Kim, MD, Principal Investigator — National Health Insurance Service Ilsan Hospital; Joonhyuk Kong, MD, Principal Investigator — Kangbuk Samsung Hospital; Stefan Betge, MD, Principal Investigator — Jena University Hospital; Holger Reinecke, MD, Principal Investigator — Universitätsklinikum Münster; Oliver Müller, MD, Principal Investigator — Universitätsklinik Heidelberg; Erwin Blessing, MD, Principal Investigator — Klinikum Karlsbad-Langensteinbach; Thomas Zeller, MD, Principal Investigator — Universtiäts-Herzzentrum Freiburg und Bad-Krozingen; Christine Espinola-Klein, MD, Principal Investigator — Johannes Gutenberg University Mainz
Locations (34):
- United States (15):
  - Cardiology, P. C. and Center for Therapeutic Angiogenesis, Birmingham, Alabama
  - Tampa Bay Medical Research, Clearwater, Florida
  - Florida Researc Network, LLC, Gainesville, Florida
  - DMI Research, Pinellas Park, Florida
  - Dr. Nadarajah Janaki, Evans, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Kentucky Research Foundation, Lexington, Kentucky
  - Cardiovascular Division, MMC, University of Minnesota, Minneapolis, Minnesota
  - Cardiovascular Institute, Mount Sinai School of Medicine, New York, New York
  - Duke University, Durham, North Carolina
  - Dr. Mohler Emile, Philadelphia, Pennsylvania
  - Omega Medical Center, Warwick, Rhode Island
  - Turkey Creek Medical Center, Knoxville, Tennessee
  - Clinical Trials of Texas, San Antonio, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Germany (9):
  - Universtiäts-Herzzentrum Freiburg und Bad-Krozingen, Bad Krozingen
  - Franziskus-Krankenhaus, Berlin
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - ASKLEPIOS Klinik St. Georg, Hamburg
  - Universitätsklinik Heidelberg, Heidelberg
  - Universitätsklinikum Jena, Jena
  - SRH Klinikum Karlsbad-Langensteinbach, Karlsbad
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsklinikum Münster, Münster
- Israel (2):
  - "Mor" Instituite, Horev M.C, Haifa
  - Edith Wolson Medical Center, Holon
- South Korea (8):
  - Dong-A University Hospital, Seo-gu, Busan
  - Korea University Ansan Hospital, Ansan, Gyeonggi-do
  - National Health Insurance Service Ilsan Hospital, Ilsandong-gu, Goyang-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Dr. Sungwon Chung, Busan
  - Dr. Weonyong Lee, Gyeonggi-do
  - Dr. Changyoung Lim, Gyeonggi-do
  - Kangbuk Samsung Medical Center, Seoul